CLINICAL TRIAL: NCT05473507
Title: Basal Cell Carcinoma Follow Up Study. A Prospective Study
Brief Title: A Study of Observation and Follow-up in People With Basal Cell Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-007
Record Dates: First submitted 2022-07-15; First posted 2022-07-26 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal Cell Carcinoma; Memorial Sloan Kettering Cancer Center; 21-007
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant with Basal Cell Carcinoma/BCC: Participants have been diagnosed with at least 1 Basal Cell Carcinoma/BCC based on clinical, dermoscopy, RCM (reflectance confocal microscopy) and OCT (optical coherence tomography)
  Interventions: Diagnostic Test: Digital Dermoscopy; Diagnostic Test: Reflectance confocal microscopy (RCM); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Dermtech tape-stripping; Diagnostic Test: Total Skin Examinations

INTERVENTIONS:
Diagnostic Test: Digital Dermoscopy — Digital Dermoscopy will be performed every 3 months.
Diagnostic Test: Reflectance confocal microscopy (RCM) — Reflectance confocal microscopy (RCM) will be performed every 3 months.
Diagnostic Test: Optical coherence tomography (OCT) — Optical coherence tomography (OCT) will be performed every 3 months.
Diagnostic Test: Dermtech tape-stripping — Dermtech tape-stripping for genetic analysiswill be performed every 6 months.
Diagnostic Test: Total Skin Examinations — Total Skin Examinations will be performed every 12 months.

SUMMARY:
The purpose of this study is to find out more about how Basal Cell Carcimonas/BCCs grow and to learn more effective ways to monitor and treat these common cancers. This study will not provide any type of treatment for the participants' cancer; it is a 3-year observational study to monitor participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Diagnosed with at least 1 BCC based on clinical, dermoscopy, RCM and OCT
* Patients with BCCs that have a diameter smaller or equal to 1.5cm, allowing for 0.5cm growth before reaching the cutoff for stage 2 BCC, which would require removal of the BCC.
* Patients with BCCs that have a depth smaller or equal to 0.6mm, to allow for tumor growth of 0.2mm before reaching the depth limitation of OCT imaging (0.8mm)
* Treatment naiive lesions
* Ability to sign informed consent

Exclusion Criteria:

* Immunosuppressed patients, such as those with a primary immunodeficiency caused by a genetic abnormality and a secondary immunodeficiency caused by AIDS, cancer, chemotherapy and other immunomodulating drugs, solid organ transplant recipitents, CLL, aspelenia, and pregnancy).
* Patients with cancer genetic syndromes that increase risk of BCC (such as basal cell nevus syndrome, xeroderma pigmentosum, epidermolysis bulosa, oculocutaneous albinism, bazex-dupre-christol syndrome, rothmund-thomson syndrome, and epidermodysplasia verruciformis).
* Patients with BCCs that are clinically suspected as high risk histopathologic subtypes, i.e. indented or sclerotic lesions that are suspected as morpheaform or infiltrative BCCs.
* Patients with BCCs that have a diameter larger than 1.5cm\
* Patients with BCCs that have a depth greater than 0.6mm
* Patients with BCCs in high risk locations, i.e. "H" area of the face. (is located in the mid-face at the site of the embryologic fusion plates and is generally believed to be associated with more aggressive skin cancers).
* Patients with BCCs on locations that may compromise an organ function should the tumor enlarge (for example, eyelid).
* Tumor located on a site that precludes attachment of the RCM device or inability to tolerate imaging procedure (i.e. remain relatively still for multiple short durations of 3- 4 minutes over a total time of 20-30 minutes)
* Lesions that previously received therapeutic intervention
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with at least 1 BCC eligible for the study will be recruited from the Memorial Sloan Kettering Dermatology sites at the Manhattan and Hauppauge clinics. Only 1 of the participant's BCCs will be selected for inclusion in the study. All patients 18 years of age or older who have been diagnosed with BCC will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Basal Cell Carcinoma growth from Baseline | 3 years
  To adequately measure the growth dynamics of tumors, several imaging modalities will be employed. Longest dimension (millimeters) of the lesion from clinical imaging will be the primary measurement of horizontal extent of the lesion. Maximum lesion depth (millimeters) from OCT imaging will be the primary measured of vertical extension.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 3 years
  To evaluate the feasibility of active follow-up of BCC as a way of managing BCC.

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Marghoob, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org